CLINICAL TRIAL: NCT04163978
Title: Phase 2 Trial to Evaluate Safety & Efficacy of Topical Nitric Oxide Releasing Sinus Irrigation (NOSi) as Compared to Budesonide-Saline (Control) in the Management of Biofilm-Associated Recalcitrant Chronic Rhinosinusitis (RCRS)
Brief Title: Nitric Oxide Releasing Sinus Irrigation (NOSi) to Treat Recalcitrant Chronic Rhinosinusitis (RCRS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanotize Research and Development corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOSi-CTP-02
Record Dates: First submitted 2019-10-31; First posted 2019-11-15 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-04

CONDITIONS: Chronic Sinusitis
Keywords: nitric oxide, sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Nitric Oxide; Therapeutics; Budesonide

STUDY DESIGN:
Intervention Model Description: Prospective double-blind, randomized, controlled, parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Investigators, and Assessors/Adjudicators will be blinded to assignment. One unblinded research coordinator at the site to complete the initial and interim dose administration and IMP reconciliation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric oxide releasing solution (NOSi) (Experimental): DailyTopical sinus irrigation delivery of 240mL NOSi
  Interventions: Drug: Nitric Oxide
- Budesonide -saline (Active Comparator): Daily Topical sinus irrigation delivery of 240 mL of 1 mg Budesonide-saline
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Nitric Oxide — in situ 240mL nitric oxide releasing sinus irrigation solution
  Other Names: Treatment
  Arms: Nitric oxide releasing solution (NOSi)
Drug: Budesonide — Saline based sinus irrigation 1mg Budesinide solution
  Other Names: Comparator
  Arms: Budesonide -saline

SUMMARY:
This a single center, randomized controlled trial to evaluate safety & efficacy of topical nitric oxide releasing sinus irrigation (NOSi) as compared to budesonide-Saline (Control) in the management of biofilm-associated recalcitrant chronic rhinosinusitis (RCRS). It is hypothesized that a daily treatment of NOSi over a 6-week period will be safe and effective at reducing clinical symptoms associated with RCRS.

DETAILED DESCRIPTION:
This is a prospective, single center, Phase 2, double-blinded, randomized, controlled, parallel group trial study. Up to fifty-four (54) participants will be enrolled (based on power analysis based on outcomes from a previous dose-tolerance study. Screening data will be reviewed to determine participant eligibility. Participants who meet all inclusion criteria and none of the exclusion criteria will be entered into the study and randomized in to the Investigational Medicinal Product (IMP) or Non Investigational Medicinal Product (NIMP) at a 2:1 ratio (NOSi:Budesonide). Each participant will be managed as an outpatient for the 42 days of the study. Participants will be administered NOSi or budesonide in saline by self-administration, at home, as a sinus irrigation to their nasopharynx and sinuses once a day. Participants will be asked to return to the clinic for evaluations on Day 21(±2), Day 43(±2) and Day 63 (±2) following the start of study interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained from the participant prior to entering the study.
2. Must be ≥ 19 years of age unless local laws dictate otherwise
3. English speaking
4. Willing and able to return to the study site for protocol required visits.
5. Documented diagnosis of chronic sinusitis with biofilm after a treatment of at least 3 months of a combination of well executed sinus surgery, regular irrigation with topical steroids or a mucosal atomization device and surfactants and at least one course of culture directed oral antibiotics
6. Persistent or worsening symptoms within 30 days of wash-in with budesonide. Specifically, documented by two SNOT-22 scores greater than or equal to 20 indicating stable (within 9 points) or worsening symptoms. SNOT-22 evaluations must be at least 7 days and no more than 30 days apart. Second SNOT-22 must be used as baseline.
7. Participant has been on a stable course of only Pulmicort and saline irrigation for a minimum of 30 days prior to randomization
8. Must be willing to use an adequate and documented form of contraception (or abstinence) from the time of the first dose with the IMP until after the last dose of IMP

Exclusion Criteria:

1. Presence of prior history of sinonasal tumors
2. Isolated sphenoid sinusitis or other sinus cavities that are not accessible to a nasal/sinus rinse as done by the patient in the head forward position
3. Autoimmune diseases affecting the upper airway eg Systemic lupus erythematosus, Sjögren's syndrome, systemic sclerosis etc
4. Immuno-compromised patients, and patients with impairment in mucociliary function (e.g., cystic fibrosis, Kartagener syndrome)
5. Severe underlying disease with anticipated survival less than 6 months
6. Females who are pregnant, breastfeeding, or plan to become pregnant during the course of the study up to 1 weeks after the last dose/study visit
7. Has used any investigational drug(s) within 30 days preceding randomization visit (Day 1);
8. Suffers from a condition, which, in the opinion of the medical investigator, would compromise their safety and / or their adherence to the study protocol
9. Systemic antibiotics, corticosteroids or antifungals within 30 days of randomization
10. Intranasal or irrigation with antibiotics, antifungals or antiseptics or any other sinusitis treatment other than Pulmicort within 30 days of randomization
11. Has a family member living in the same household, also enrolled or planning to enroll in this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of NOSi compared to Budesonide on disease specific quality of life in participants with biofilm-associated recalcitrant chronic rhinosinusitis (RCRS) as measured by the Sino-Nasal Outcome Test (SNOT-22) | 42 days
  Proportion of participants experiencing a 9-point reduction in Sino-Nasal Outcome test (SNOT-22) score (0-5 scale of 22 parameters with a total maxmimum score of 110 and an increased value representing worsening of condition)
To assess the safety of NOSi compared to Budesonide on disease specific quality of life in participants with biofilm-associated recalcitrant chronic rhinosinusitis | 63 days
  Severity and frequency of adverse events as well as clinically significant Changes in laboratory findings, vital signs, histology, olfaction, and methemoglobin levels.

SECONDARY OUTCOMES:
To evaluate the efficacy of NOSi compared to Budesonide on the reduction of Modified Lund-Kennedy Scores (MLK) | Days 21, 42, 63
  Mean change in MLK score as compared to control (Scale of 0-2 for 6 locations on each side (maximum total score 24); increase represents worsening
To evaluate the efficacy of NOSi compared to Budesonide on quality of life improvements (EQ-5D-5L); | Days 21, 42, 63
  Mean change in EQ-5D-5L index score as compared to control (Scale 0-100; increase indicates worsening)
To evaluate the efficacy of NOSi compared to Budesonide on the density of pathogens | Days 21, 42, 63
  Mean change in pathogen density compared to control; (log10 cfu/g)
To evaluate the efficacy of NOSi compared to Budesonide on cilia functionality | Days 43 & 63
  Proportion of participants with functional cilia which is known to be denuded by biofilm as determined by the saccharin test compared to control
To evaluate the efficacy of NOSi compared to Budesonide on biofilm elimination | Days 43 & 63
  Proportion of participants with biofilm elimination compared to control

CONTACTS AND LOCATIONS:
Overall Officials: Amin Javer, MD, Principal Investigator — St. Paul's Hospital
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No